CLINICAL TRIAL: NCT05854849
Title: A Multicenter, Phase 3 Clinical Trial of Gemcitabine and Camrelizumab Plus Apatinib Versus Cisplatin in First-line Treatment of Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Gemcitabine and Camrelizumab Plus Apatinib Versus Cisplatin in First-line Treatment of RM-NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2023-GAPvsGPP
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; PD-1; metastatic
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis | interventions — camrelizumab; Gemcitabine; Cisplatin; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAP (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Gemcitabine; Drug: Apatinib
- GPP (Active Comparator)
  Interventions: Drug: Camrelizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Camrelizumab — 200mg, D1, Q3W, iv drip.
Drug: Gemcitabine — 1000mg/m2, Day 1 and Day 8, Q3W, iv drip, maximum 6 cycles.
Drug: Cisplatin — 80 mg/m2, D1, Q3W, iv drip, maximum 6 cycles.
  Arms: GPP
Drug: Apatinib — 250mg, PO, QD
  Arms: GAP

SUMMARY:
This study aims to explore a new, more effective and tolerable treatment regimen for patients with advanced recurrent/metastatic nasopharyngeal carcinoma. Specifically, we plan to conduct a phase III randomized controlled clinical trial based on the standard treatment of "GP + PD-1 mAb", replacing cisplatin with apatinib to achieve "platinum-free" therapy and reduce toxicity. In addition, we will investigate the efficacy of using apatinib in combination with PD-1 mAb compared to PD-1 mAb monotherapy to further improve treatment outcomes. The ultimate goal is to provide a new and reliable treatment modality for patients with advanced recurrent/metastatic nasopharyngeal carcinoma and guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; 18-70 years of age;
2. Had histopathologically confirmed nonkeratinizing recurrent/metastatic NPC (AJCC, 8th; the metastatic tissue biopsy is preferred, not necessary; locoregional recurrent lesion unfit for local treatment).
3. Did not receive any systemic treatment for recurrent and metastatic lesions. (Previous radiotherapy, induction chemotherapy, concurrent chemoradiotherapy, or adjuvant chemotherapy should have been completed at least 6 months prior to treatment)
4. ECOG performance status of 0 or 1.
5. Subjects enrolled must have measurable lesion(s) according to response evaluation criteria in solid (RECIST) v1.1.
6. Adequate organ function assessed by laboratory parameters during the screening period
7. Life expectancy more than 12 weeks.
8. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Patients with a high risk of nasopharyngeal necrosis: ① Patients with recurrent stage T3-4 received two courses of radiotherapy before enrollment, or received nasopharyngeal radiotherapy within 1 year before enrollment; ② Patients with recurrent T1-2 stage had received two courses of nasopharyngeal radiotherapy and the last radiotherapy within 1 year before enrollment.
2. Patients with other malignancies (except for cervical cancer, basal cell carcinoma or squamous cell carcinoma of the skin, localized prostate cancer, and ductal carcinoma in situ who have undergone curative treatment).
3. Special attention: Patients with active bleeding, ulcers, bowel perforations, and major surgery within 30 days; tumors in close proximity to the internal carotid artery or other major vessels, and those at risk of major bleeding. Patients with or previous with serious hemorrhage (bleeding >30 ml within 3 months), haemoptysis (> 5 ml within 4 weeks) of thromboembolic events within 12 months (including stroke events and/or transient ischemic attack).
4. Patients with hypertension who cannot be reduced to the normal range by antihypertensive drug treatment (systolic blood pressure > 140 mmHg/diastolic blood pressure > 90 mmHg), patients with ≥ grade II coronary heart disease, arrhythmia (including QTc interval prolongation > 450 ms in men and > 470 ms in women) and cardiac insufficiency.
5. Patients with known or suspected autoimmune diseases including dementia and seizures.
6. Multiple factors affecting the absorption of oral medications (e.g., dysphagia, chronic diarrhea, and bowel obstruction).
7. An excessive dose of glucocorticoids given within 4 weeks before enrollment.
8. Complications requiring long-term use of immunosuppressive drugs or systemic or local use of immunosuppressive-dose corticosteroids.
9. HIV positive; HBsAg positive and HBV DNA copy number positive (quantitative detection ≥ 1000 cps/ml); chronic hepatitis C with blood screening positive (HCV antibody positive).
10. Women of childbearing age with a positive pregnancy test and lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  the time from treatment initiation to disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 2 years
  the survival time until death from any cause
Objective response rate | 2 years
  the proportion of patients with complete response (CR) or partial response (PR) according to RECIST v1.1
Disease control rate | 2 years
  the proportion of patients who achieved CR, PR, or stable disease
Duration of response | 2 years
  the time from the first evidence of response to disease progression or death
Safety evaluation | 2 years
  incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China